CLINICAL TRIAL: NCT01046812
Title: Halitosis Devised Questionnaire Evaluating a New Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Head & Neck Institute (Other)
Responsible Party: Victor Kizhner, SLLR
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLR 09-141
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2009-12

CONDITIONS: Halitosis
Keywords: questionnaire; halitosis; caphosol; Quality of life questionnaire assessing halitosis
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Caphosol — Caphosol 2-4 times daily oral rinse for two weeks duration minimum up to one month.

SUMMARY:
The investigators propose a novel assessment of oral malodor (halitosis) by a quality of life (QOL) questionnaire designed specifically for halitosis and a new treatment for halitosis by improvement of mouth dryness.

DETAILED DESCRIPTION:
Halitosis is a common symptom which can affect people of all ages. It may decrease self confidence and social interactions. Oral halitosos is the consequence of microbial (mainly Gram negative bacteria) breakdown of food debris, cells, saliva, and blood. The agents that give rise to halitosis include especially the volatile sulphur compounds (VSC), diamines, and short chain fatty acids of which only the VSC can be detected in the clinical setting, making the detection of halitosis often very hard. The most common cause for oral halitosis is poor oral hygiene due to gingivitis or periodontitis. Other causes include bacterial accumulation on the posterior tongue, tonsillitis and others. Dry mouth has been implicated as a potential cause in halitosis.

Due to the lack of quantitative objective measuring to the severity of halitosis and especially in the face of the subjective nature of halitosis as occurs commonly a subjectively measurement is necessary. As no current QOL exists for measurement of halitosis formulation of such a questionnaire can enable a measurement of subjective halitosis with change observed over time or with intervention.

We intend to treat halitosis with a novel approach targeting mouth dryness- when other factors were ruled out by measuring outcome on the halitosis questionnaire.

We will treat mouth dryness with Caphosol- a solution indicated for mouth dryness acting only locally after mouth washing. As this is a supersaturated phosphate solution of a mineral not alien to the body side effects are practically negligible.

Quality of life (QOL) questionnaires (such as SNOT20- sinonasal outcome test) are common in medicine, however no such questionnaire exists for halitosis. We devised a specific QOL questionnaire for halitosis. This questionnaire consists of 20 questions covering functional limitation, physical discomfort, psychological discomfort, physical disability and social disability. The answers will be based on a common scale of 5 answers depending on the severity and ranging from a never bothering symptom to a symptom which as worse as can be. Formulation of this a questionnaire can assist in measuring subjective halitosis with change observed over time or with intervention.

Treating halitosis is a challenge due to the multitude of factors. However, some treatments, mainly in the form of nasal saline irrigation or oral solutions chlorine based or triclosan exist. Mouth dryness, although implicated as a factor, has not been targeted yet. Improving salivary flow may reduce the stasis of saliva thus reducing the concentration of proteins that bacteria dwell on as well as a better degradation of oral food debris.

Caphosol is a topical oral agent of supersaturated calcium phosphate rinse indicated for dry mouth that has been clinically proven to shorten the duration and severity of mucositis and relieve dry mouth when used with fluoride. Caphosol is indicated for dryness of the mouth or throat (hyposalivation, xerostomia), regardless of the cause and regardless of whether the conditions are temporary or permanent. Caphosol is also indicated as an adjunct to standard oral care in treating the mucositis that may be caused by radiation or high dose chemotherapy. It has an extremely high safety profile as these salts are not alien to the body, thus if swallowed accidentally, no adverse effects are expected. No known drug interactions exist.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of halitosis
* Patients over 18
* Patients with dry mouth as seen on physical examinations
* Patients that may be suffering from Sjogren's syndrome will be screened by SSB/La blood test.

Exclusion Criteria:

* Patients without any other noted causes contributing to halitosis.
* Patients restricted to a low sodium diet without specific permission from the treating physician.
* Patients not wishing to participate in the study will be asked to fill the questionnaire regardless

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of Caphosol in treating Halitosis | 1 month

SECONDARY OUTCOMES:
Confirmation of QOL questionnaire as tool measuring the burden of halitosis | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- New York Head & Neck Institute offices, New York, New York, United States

REFERENCES:
- [Background] Porter SR, Scully C. Oral malodour (halitosis). BMJ. 2006 Sep 23;333(7569):632-5. doi: 10.1136/bmj.38954.631968.AE. No abstract available. PMID 16990322
- [Background] Koshimune S, Awano S, Gohara K, Kurihara E, Ansai T, Takehara T. Low salivary flow and volatile sulfur compounds in mouth air. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2003 Jul;96(1):38-41. doi: 10.1016/s1079-2104(03)00162-8. PMID 12847442
- See also: New York Head & Neck Institute — http://nyhni.org/
- See also: Dr.Krespi's detailed resume — http://nyhni.org/faculty/yosef_krespi/index.html